CLINICAL TRIAL: NCT03986801
Title: Impact of a Permanently Maintained Healthcare Multidisciplinary Facility Named Permanece d'Accès Aus Soins de Santé (PASS-MULTI) on Unscheduled Readmissions at 12 Months for Persons in Precarious Situations.
Brief Title: Impact of a Permanently Maintained Healthcare Multidisciplinary Facility (PASS-MULTI) on Unscheduled Readmissions at 12 Months for Persons in Precarious Situations.
Acronym: PASS-MULTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-03
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Vulnerable Patients

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized between a non-interventional group (standard management of patients according to the institution of origin) or intervention group (setting up a PASS pharmaceutical interview on the day of discharge from hospital and follow-up multidisciplinary until rights are obtained).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASS pharmaceutical interview (Experimental)
  Interventions: Other: pharmaceutical interview
- Usual management out of hospital (No Intervention)

INTERVENTIONS:
Other: pharmaceutical interview — pharmaceutical interview at the end of hospitalization
  Arms: PASS pharmaceutical interview

SUMMARY:
Created in 1998, PASS departments are mostly intrahospital structures providing primary care to vulnerable patients.

The main objective of the project will be to measure the impact of a multidisciplinary PASS benefiting from outpatient pharmaceutical interviews on the rate of unplanned rehospitalization of patients in precarious situations.

The impact of the implementation of such a device will also be measured on other indicators of major interest in the course of care of the precarious patient: average lengths of stay, emergency room, improved continuity of treatment, quality of life of the patient related to his health, medication compliance, effective accessibility to social rights, qualitative improvement in the use of care, medico-economic efficiency of the intervention compared to existing practice.

The study will be multicenter: 6 centers spread throughout France (Marseille, Paris, Nice, Toulouse, Poitiers and Bayonne).

DETAILED DESCRIPTION:
Created in 1998, PASS ( Permanence d'Accès aux Soins de Santé) departments are mostly intrahospital structures providing primary care to vulnerable patients.

This facility allows medico-social care for people in precarious situations, for a return to the common health system. However, the individual difficulties to resort to care, complicated by a system of health sometimes excluding, and the dissociation of the activity of dispensing treatments from the action of the PASS can lead to breaks of treatments, can cause pathological complications, or cause re-hospitalization. More particularly, the methods of dispensing drugs and medical devices for outpatients in precarious situations are very heterogeneous depending on the institutions and the geographical distance of the PASS or the PUI: discharge with orientation towards the PUI and PASS; dispensing via the unitcare by a doctor or social worker; discharge without medication, without orientation and only with a prescription,... Actually, in some cases, it is highlighted the question of the renewal of treatments and the rupture of these and therefore the breakdown of care.

The use of original and innovative practices, including pharmaceutical maintenance and multidisciplinary monitoring (social, medical and pharmaceutical) until the social rights are obtained, is therefore necessary to promote a reliable and effective system for the care of precarious patients, but also to reassure the patient in his care pathway.

The main objective of the project will be to measure the impact of a multidisciplinary PASS facility, integrating pharmaceutical interviews, for outpatient, on the rate of unscheduled rehospitalization of patients in precarious situations.

The impact of the implementation of such a facility will also be measured on other indicators of major interest in the care pathway of the precarious patient: average lengths of stay, emergency room, improved continuity of treatment, quality of life of the patient related to his health, medication compliance, effective accessibility to social rights, qualitative improvement in the use of care, medico-economic efficiency of the intervention compared to existing practice.

Eligible patients will be randomized between a non-interventional group (standard management of patients according to hospital) or interventional group (setting up a PASS pharmaceutical interview on the day of discharge from hospital and multidisciplinary follow-up until social rights are obtained).

The intervention will consist in the overall medico-social care of the patient in precarious situation by the Multidisciplinary PASS facility, at discharge, including a specialized pharmaceutical interview (PI) while dispensing the treatments; then monthly PI, concomitantly with medical consultations and social follow-up until the end of the study or opening of social rights.

In the non-interventional group, the discharge of the precarious patient will be implemented according to the usual methods of each hospital: the unitcare will have the mission of refering the patient towards the medico-social PASS, and of ensure that the patient is in possession of the necessary documents for the dispensing of the treatments; but this one will not benefit from PI.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Informed consent form signed by the subject
* Inpatient hospitalized for over 24 hours
* Precarious socioeconomic conditions (EPICES Score 30)
* Incomplete social security cover

Exclusion Criteria:

* Children
* Refusal of consent
* Outpatients
* No precarious socioeconomic conditions (EPICES Score Under 30)
* Complete social security cover (AMU, CMUc, ACS, ALD)
* Majors in tutorship or guardianship, pregnant women and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1858 (Estimated)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2020-09-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
The number of unscheduled hospitalizations | 12th month of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France